CLINICAL TRIAL: NCT04281446
Title: Mapping the Physical Performance of Women From Endogenous Ovarian Cycles at Different Stages of the Menstrual Cycle, and the Respective Influence of Photobiomodulation Therapy
Brief Title: Physical Performance of Women at Different Stages of the Menstrual Cycle, and Photobiomodulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, P.h.D Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1143-7630
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Menstrual Cycle Disorder
Keywords: Menstrual cycle; Photobiomodulation therapy; Fatigue; Clinical Trial
MeSH Terms: conditions — Menstruation Disturbances; Fatigue | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The randomization and allocation of participants will be performed at beginning of the project, allocating the participants in 2 groups:
  * Endogenous ovarian cycle Photobiomodulation Group(G-FBM-CEN);
  * Endogenous ovarian cycle Sham Group (G - Sham - CEN).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization and allocation of participants will be performed by a researcher who will not have access to evaluations and data collection. The interventions will be carried out by the researcher who made the allocation, and data collection by a second researcher, who is blinded to the allocation of the participants.
  Participants will not know about their allocation during the collection process and during the intervention they will wear a mask covering their eyes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-FBM-CEN (Experimental): Photobiomodulation application in women of endogenous cycle. Antares® equipment (IBRAMED, Amparo-SP, Brazil) will be used, by means of a cluster, with two wavelengths (13 LEDs of 630 nm, 300 mW + 13 LEDs of 850 nm, 500 mW), being its area of 80 cm² contact, acting 180 J of energy being applied at 15 points on each thigh - 9 in the anterior region and 6 in the posterior region, in addition to 2 points in the gastrocnemius.
  Interventions: Device: Photobiomodulation
- G - Sham - CEN (Sham Comparator): Sham Photobiomodulation (disabled) application in women of endogenous cycle.
  The procedure and equipment will be the same as for the experimental groups, however no dosage will be applied:
  Antares® equipment (IBRAMED, Amparo-SP, Brazil) will be used, by means of a cluster, with two wavelengths (13 LEDs of 630 nm, 300 mW + 13 LEDs of 850 nm, 500 mW), being its area of 80 cm² contact, with 0 J of energy being applied at 15 points on each thigh - 9 in the anterior region and 6 in the posterior region, in addition to 2 points in the gastrocnemius.
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Application of light at specific wavelength for interaction with biological tissue

SUMMARY:
Hormonal fluctuations present during the ovarian cycle may have a strong influence on physiological and psychological aspects on physical performance in women. The aspects surrounding performance and ovarian cycles in women during different phases of the cycle, are still current and should be debated in the literature, as the available evidence has conflicting results. In addition to the above, new ergogenic methods have been studied to improve the sports scenario in different populations. Research on the use of ergogenic electrophysical resources so that hormonal effects may possibly be mitigated, allowing women to use this resource and improving their physical performance is still scarce in the current literature.

DETAILED DESCRIPTION:
Objective: To evaluate the physical performance of women during different phases of the ovarian cycle and the influence of photobiomodulation therapy in this setting. Methods: The research will be conducted in two subprojects - Subproject I is a cross-sectional study. Initially the participants will be evaluated in two phases separately, being the first and second day within the ovarian cycle in the follicular phase (FF) and the third and fourth day in the luteal phase (FL). The aspects of body composition, body water volume and skin temperature by infrared thermography will be evaluated, and the physical performance evaluation will be constituted by the evaluation of the muscular performance by isokinetic dynamometer, and by a treadmill supramaximal effort test. , together with analysis of VO2max and blood lactate levels. Subproject II is a double-blind placebo-controlled randomized clinical trial. After completion of subproject I, during the next ovarian cycle within the participants will return to conduct the second part of the study, which will analyze the influence of photobiomodulation therapy on the physical performance of women within their menstrual cycle, related to low hormone rate ( FF). 200 J of energy will be applied before each evaluation, which is muscle performance and endurance. The tests will be performed in the same order, following the same protocol in both phases of the study. For data analysis, a normality test will be used to verify the distribution and statistical tests consistent with the appropriate intra and intergroup comparisons, being considered two factors in the comparisons, time and group. A significance level of 5% will be adopted. The effect size will be calculated by Cohens'd.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 to 35 years
* Healthy
* Physically Active (150 min / week)

Exclusion Criteria:

* Eating disorders;
* Hormonal disorders;
* Amenorrhea;
* Pregnancy;
* Polycystic ovary;
* Endometriosis;
* Tumors;
* Musculoskeletal injury in the last 6 months;
* Cardiorespiratory disease;
* Use of alcohol and illegal drugs during the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Fatigue Strength | 20 minutes
  Distance traveled during incremental testing (km)

SECONDARY OUTCOMES:
Muscle Performance | 20 minutes
  Quantitative assessment of muscle performance performed by isokinetic dynamometer (N/m; W, %)
Subjective Perception of Effort | 20 minutes
  Modified 10-point Borg scale
  The scale assesses the level of effort, with 0 being no effort and 10 being the maximum physical effort.
Ventilatory variables | 20 minutes
  VO2máx (ml.kg-1.min-1)
Lactate | 20 minutes
  Lactate threshold (iLL) and anaerobic threshold (iLAN) (mmol/L)
Body Temperature | 15 minutes
  Thermographic evaluation (°C)
Body water level | 10 minutes
  Bioimpedance Evaluation (%)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela de Carvalho, Ms., Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Rinaldo Roberto de Jesus Guirro, Ribeirão Preto, São Paulo
  - Universidade de São Paulo, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No